CLINICAL TRIAL: NCT01247103
Title: A Phase 1, Single-centre Randomised, Double-Blind, Placebo-Controlled, Single and Multiple Dose, Parallel-group Study to Determine the Safety, Tolerability, and Pharmacokinetics of AZD4316 in Healthy Volunteers
Brief Title: Assessment of the Safety and Pharmacokinetics of Single and Multiple Oral Doses of AZD4316 in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, Arrow Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3340C00002
Record Dates: First submitted 2010-11-16; First posted 2010-11-24 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers; safety; tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Part A: single ascending dose (Placebo Comparator): AZD4316: single oral dose, with 1 group with/without food
  Interventions: Drug: AZD4316; Other: Placebo
- Part B: multiple ascending dose (Placebo Comparator): AZD4316: multiple oral doses
  Interventions: Drug: AZD4316; Other: Placebo

INTERVENTIONS:
Drug: AZD4316 — Single oral doses of AZD4316 suspension in the fasted state. In one group in Part A, subjects will receive a second dose of AZD4316 in the fed state (within 30 min after receiving a high fat breakfast)
  Arms: Part A: single ascending dose
Drug: AZD4316 — Multiple oral doses of AZD4316 suspension. It's planned that doses will be administered in the fasted state, however, if in Part A it's shown that food increases absorption of AZD4316, then doses will be administered after a meal.
  Arms: Part B: multiple ascending dose
Other: Placebo — Placebo to match AZD4316

SUMMARY:
The purpose of the study is to assess the safety, tolerability and pharmacokinetics of AZD4316 following oral administration of single and multiple doses to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 50 years with suitable veins for cannulation or repeated venepuncture.
* Female subjects must not be pregnant, must not be lactating and must be of non-child-bearing potential (i.e. they must be post-menopausal or surgically sterile)
* Male subjects should be willing to use barrier contraception i.e. condoms and spermicide, from the day of dosing until at least 3 months after dosing with the investigational product
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Subjects who are healthy as determined by pre study medical history, physical examination, 12-Lead ECG

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG, including changes that may interfere with the interpretation of QTcF interval changes.
* Current smokers, those who have smoked or used nicotine products within the previous three months.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4316.
* Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | from screening period to follow-up
Assesment of vital signs (blood pressure, pulse and temperature) | from screening period to follow-up
  Frequent assessments will be made for each subject from the screening period to follow up
Assessment of laboratory variables and physical examinations | from screening period to follow-up
  Frequent assessments will be made for each subject from the screening period to follow up
Assessment of Electrocardiogram (ECG) variables | from screening period to follow-up
  Frequent assessments will be made for each subject from the screening period to follow up

SECONDARY OUTCOMES:
Pharmacokinetic variables of AZD4316 by assessment of drug concentrations in plasma and urine | Serial blood samples and urine collection for PK evaluation throughout the period of admission and up to the time of the follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Dr Dereck Tait, Study Director — Arrow Therapeutics; Dr Darren Wilbraham, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, London, United Kingdom